CLINICAL TRIAL: NCT06733064
Title: Effective Prevention of Osteoporosis Through Rehabilitation and Training
Brief Title: Strenght Training in Osteoporosis Prevention
Acronym: SPORT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mateusz Karnia (Other)
Responsible Party: Sponsor-Investigator, Mateusz Karnia, Principal Investigator, University of Gdansk
Organization: University of Gdansk (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Komisja Bioetyczna-47/23; NdS-II/SP/0449/2024/0 (Other Grant/Funding Number: The Polish Ministry of Science and Higher Education)
Record Dates: First submitted 2024-11-08; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Osteopenia or Osteoporosis
Keywords: strenght training; vitamin d3; osteoporosis; osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D3 supplementation (Experimental): Group receiving vitamin D3 at a dose of 4000 IU / day
  Interventions: Dietary Supplement: Supplementation of vitamin D3
- Placebo supplementation (Placebo Comparator): Vegetable oil as a placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Supplementation of vitamin D3 — Supplementation of vitamin d3 at a dose of 4000 iu / day
  Arms: Vitamin D3 supplementation
Dietary Supplement: Placebo — Vegetable oil as a placebo
  Arms: Placebo supplementation

SUMMARY:
The study involves 120 women over the age of 50.

All participants in the study take part in high-intensity strength training for 10 months.

In addition, half of the participants receive vitamin D3 at a dose of 4,000 IU/day.

The investigators hypothesize that training combined with vitamin D3 supplementation will be more effective in preventing osteoporosis than training alone.

ELIGIBILITY:
Inclusion Criteria:

* age over 50
* female

Exclusion Criteria:

* ongoing cancer,
* unstabilized cardiovascular disease,
* cognitive disorders,
* radiological treatment in the last 12 months,
* other contraindications to undertaking high-intensity strength training,
* diseases affecting the skeleton such as: Paget's disease, type I diabetes mellitus,
* taking medications affecting skeletal conditions including: long-term therapy with corticosteroids, thiazides, antiretroviral drugs,
* contraindications to taking vitamin D including: hypercalcemia, nephrolithiasis, sarcoidosis, lack of cholecalciferol hydroxylase activity in the liver and kidneys.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density | Measured at 3 time points: before the experiment, after 10 months of training, and at 6 months after the end of training and supplementation.
  Test to determine bone mineral density by densitometry.

SECONDARY OUTCOMES:
Vitamin D metabolites level | Measured at 4 time points: before the experiment, after 5 and 10 months of training, and at 6 months after the end of training and supplementation.
  Measurement evaluating the levels of selected vitamin D3 metabolites by LC-MS.

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz Karnia, PhD, Principal Investigator — University of Gdansk
Locations (2):
- Poland (2):
  - University of Gdańsk, Faculty of Biology, Gdansk, Pomeranian Voivodeship
  - University of Gdańsk, Faculty of Biology, Gdansk

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://projekt-sport.ug.edu.pl